CLINICAL TRIAL: NCT00038623
Title: A Phase II Study Of Yttrium-ibritumomab (Zevalin) For the Treatment Of Patients With Relapsed And Refractory Mantle Cell Lymphoma
Brief Title: Study Of Yttrium-ibritumomab (Zevalin) For the Treatment Of Patients With Relapsed And Refractory Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID01-541
Record Dates: First submitted 2002-06-03; First posted 2002-06-04 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-10

CONDITIONS: Lymphoma, Mantle-Cell
Keywords: Relapsed/Refractory Mantle Cell Lymphoma; Yttrium-Ibritumomab; Zevalin
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — ibritumomab tiuxetan; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Yttrium-ibritumomab (Zevalin) (Experimental): After Rituximab infusion (250 mg/m^2 intravenous) on Day 1, 111^In Zevalin on Day 1 followed by two whole body imaging performed on Day 1 then Day 2.
  Interventions: Drug: Yttrium-ibritumomab (Zevalin); Drug: Rituximab

INTERVENTIONS:
Drug: Yttrium-ibritumomab (Zevalin) — After Rituximab infusion, 111^In Zevalin on Day 1 followed by two whole body imaging performed on Day 1 then Day 2.
  Other Names: 90-Yttrium-ibritumomab; Zevalin; IDEC-Y2B8; Ibritumomab; Ibritumomab tiuxetan
Drug: Rituximab — 250 mg/m^2 in the vein over 6 to 8 hours on Day 1.
  Other Names: Rituxan

SUMMARY:
Study of Yttrium-ibritumomab (Zevalin) For the treatment of Patients with Relapsed & Refractory Mantle Cell Lymphoma

DETAILED DESCRIPTION:
Mantle cell lymphoma cell express a protein called CD20. Ibritumomab tiuxetan is an antibody targeted against CD20, which carries a radioactive material called 90-Yttrium. The radioactivity will be delivered to the cancer cells by the antibody will help killing the mantle cell lymphoma cells. Before treatment starts, patients will have a physical exam, including blood and urine test. Patients will have a chest x-ray and CT scans of the abdomen and pelvis. Bone marrow samples will be taken with a large needle. A cardiogram (EKG) will be performed before therapy and after 1 and 3 months of therapy.

Patients in this study will receive one dose of rituximab in the vein over 6 to 8 hours on the first day of treatment. This will be followed by an infusion of antibody labeled with radioactive indium, which will allow imaging of the tumor sites and normal tissue site that will bind the antibody.

Imaging will be performed twice in the nuclear medicine department of Day 1, and once on either Day 2 or 3. On day 8 (7 days after the first dose of rituximab), patients will receive a second dose of rituximab. This will immediately be followed by a dose of Ibritumomab tiuxetan given by vein over ten minutes. Patients will receive diphenhydramine (Benadryl) by vein and mouth and acetaminophen (Tylenol) by mouth before each dose of rituximab. This is done to prevent fever and chills. All treatments will be given in an outpatient setting.

Blood test will be taken weekly during the first 3 months, the every 3 months for 1 year, and then every 6 months for 3 years. CT scans, x-rays, and bone marrow biopsies will be repeated if needed after 3 months of therapy and every 3 months for 1 years, then every 6 months for 3 years. If tumors do not shrink after 3 months of therapy or increase in size, patients will be offered a different treatment.

This is an investigational study. Up to 35 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed, relapsed or refractory mantle cell lymphoma requiring treatment.
2. No anti-cancer therapy for three weeks (6 weeks if rituximab, nitrosurea, or Mitomycin C) prior to study initiation, and fully recovered from all toxicities associated with prior surgery, radiation treatments, chemotherapy, or immunotherapy.
3. An IRB-approved signed informed consent.
4. Age greater or equal to 18 years.
5. Expected survival greater than or equal to 3 months.
6. Pre-study performance status of 0, 1, or 2 according to the World Health Organizations (WHO) criteria.
7. Acceptable hematologic status within two weeks prior to patient registration, including: Absolute neutrophil count (segmented neutrophils = bands * total White Blood Count (WBC)) greater than or equal to 1,500/mm^3; Platelets greater than or equal to 1000,000/mm^3.
8. Female patients who are not pregnant or lactating.
9. Men and women of reproductive potential who are following accepted birth control methods (as determined by the treating physician, however abstinence is not an acceptable method).
10. Patients previously on investigational Phase II anti-cancer drugs if no long-term toxicity is expected, and the patient has been off the drug for eight or more weeks with no significant post treatment toxicities observed.
11. Patients determined to have less than 25% bone marrow involvement with mantle cell lymphoma within six weeks of registration. Measurement to be determined by bilateral bone marrow biopsies. This criteria must be strictly met for adequate patient safety.

Exclusion Criteria:

1. Prior autologous or allogeneic bone marrow transplantation (ABMT) or peripheral blood stem cell (PBSC) rescue therapy.
2. Prior radioimmunotherapy.
3. Presence of Central Nervous System (CNS) lymphoma.
4. Patients with HIV or AIDS-related lymphoma.
5. Patients with pleural effusion.
6. Patients with abnormal liver function: Total bilirubin greater than 2.0mg/dL
7. Patients with abnormal renal function: serum creatinine greater than 2.0mg/dL
8. Patients who have received prior external beam radiotherapy to greater than 25% of active bone (involved field or regional).
9. Patients who have received Granulocyte colony-stimulating factor (G-CSF or GM-CSF) therapy within two weeks prior to treatment.
10. Serious nonmalignant disease or infection which, in the opinion of the investigator and/or sponsor, would compromise other protocol objectives.
11. Major surgery, other than diagnostic surgery, within four weeks.
12. Impaired bone marrow reserve as indicated by one or more of the following: a) History of failed stem cell collection. b) Platelet count less than 1000,000 cells/mm^3. c) Hypocellular bone marrow (less than 15% cellularity). d) Marked reduction in bone marrow precursors of one or more cell lines (granulocytic, megakaryocytic, erythroid).
13. Presence of leukemic phase of disease defined as peripheral blood absolute lymphocyte count of greater than 5,000/microliters.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2002-04; Primary Completion 2007-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Objective tumor response | Followed for 4 years or until disease progression
  Objective tumor response is defined as CR + CCR + PR, where CR = Complete Response, CCR = Clinical Complete Response and PR = partial response. All patients who receive any dose of Zevalin will be included in the calculation of response rate.

CONTACTS AND LOCATIONS:
Overall Officials: Anas Younes, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org